CLINICAL TRIAL: NCT04482803
Title: Feasibility Study of Targeted Biopsy of Carbon Nanoparticles Labelled Axillary Node After Neoadjuvant Systemic Therapy for Clinically Assessed Positive Axillary Lymph Node (cN+) Breast Cancer
Brief Title: Targeted Biopsy of Carbon Nanoparticles Labelled Axillary Node for CN+ Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jue Wang, Prof., The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NBC Sur001
Record Dates: First submitted 2020-07-04; First posted 2020-07-23 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Location and Biopsy of Axillary Lymph Nodes
Keywords: Breast cancer; neoadjuvant chemotherapy; Axillary lymph nodes positive; Carbon-tattooed Lymph Nodes; locating clip
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carbon nanoparticles labelled lymph nodes group (Experimental): Carbon nanoparticles suspension injection will be injected into or around the cortex of the clinically assessed positive lymph nodes before NST.
  Interventions: Drug: Carbon nanoparticles suspension injection will be injected into or around the cortex of the clinically assessed positive lymph nodes

INTERVENTIONS:
Drug: Carbon nanoparticles suspension injection will be injected into or around the cortex of the clinically assessed positive lymph nodes — Before NST, one of the clinically assesed positive lymph nodes will be subjected to ultrasound-guided CNB or FNA, and a locating clip (Ultraclip, BARD) will be placed. Meanwhile, a small amount of Kanarine (carbon nanoparticles suspension injection, 0.5ml:25mg, H20073246) will be injected into or around the cortex of the locating lymph node and other clinically assessed positive lymph nodes. Preoperative FNA will be performed again for locating clip labelled node.
  Other Names: A locating clip was placed in one of the suspected lymph nodes; Preoperative FNA will be performed again for locating clip labelled node

SUMMARY:
To explore the feasibility of target biopsy of carbon nanoparticles labelled lymph node after neoadjuvant systemic therapy for cN+ breast cancer, and evaluate whether it can accurately predict axillary lymph node status after neoadjuvant systemic therapy.

DETAILED DESCRIPTION:
Locally advanced breast cancer patients with clinical assessed positive axillary lymph node (cN+) who receive neoadjuvant systemic therapy (NST) will be enrolled in this study. Before NST, one of the suspected lymph nodes will be subjected to ultrasound-guided core needle biopsy (CNB) or fine needle aspiration (FNA), and a locating clip will be placed. Meanwhile, a small amount of Kanarine (Carbon Nanoparticles Suspension Injection) will be injected into or around the cortex of the locating lymph node as well as other positive lymph nodes. All patients will be confirmed to have axillary lymph node metastasis by pathologic or cytologic examination. After NST, FNA will be performed again for the lymph nodes labelled with previous locating clip. During the operation, the clip labelled lymph nodes were identified with carbon and sent to pathology separately. Meanwhile, the remaining carbon labelled lymph nodes were also separately examined. Axillary lymph node dissection will be performed in all patients. The detection rate of labelled lymph node will be record, and the pathological results of re-FNA of labelled lymph nodes will be compared with postoperative pathological results. Meanwhile, we will also analysis whether carbon labelled lymph node biopsy could predict the overall status of axillary lymph nodes after NST.

ELIGIBILITY:
Inclusion Criteria:

1. Female breast cancer patients who received neoadjuvant systemic chemotherapy, aged 18-70 years old, with clinically assessed positive lymph node, and the expected survival period is greater than 12 months.
2. No previous radiotherapy and chemotherapy.
3. No history of serious systemic disease.
4. KPS≥70.
5. White blood cell count> 3.5 × 10 ^ 9 / L, neutrophil count> 1.8 × 10 ^ 9 / L, platelet count> 100 × 10 ^ 9 / L, hemoglobin> 9 g / dl.
6. ALT and AST <1.5 times the upper limit of normal value, alkaline phosphatase <2.5 times the upper limit of normal value, and total bilirubin <1.5 times the upper limit of normal value.
7. Serum muscle plasma <1.5 times the upper limit of normal value.
8. No abnormal blood coagulation.
9. Women of childbearing age had a negative serum or urine pregnancy test before the start of treatment and agreed to contraception during treatment.
10. Cardiac function: two-dimensional echocardiography examination LVEF ≥ 55%.
11. Sign informed consent.

Exclusion critia:

1. Received systemic or local treatment for tumors, including chemotherapy, radiotherapy and endocrine therapy.
2. A history of malignant tumors within 5 years (except curable skin basal cell carcinoma and cervical carcinoma in situ).
3. The patient has been enrolled in other clinical trials or used other study drugs 30 days before enrollment in this study.
4. Accompanied by uncontrolled lung disease, severe infection, active gastrointestinal ulcer need treatment, coagulopathy, severe uncontrolled diabetes, connective tissue disease or bone marrow function suppression and other diseases, can not tolerate chemotherapy related treatments.
5. Two-dimensional echocardiography detection LVEF <55%.
6. Severe cardiovascular and cerebrovascular diseases within the first 6 months of randomization (eg unstable angina, chronic heart failure, uncontrollable hypertension> 150/90 mmHg, myocardial infarction or cerebrovascular accident).
7. NCI peripheral neurotoxicity grade ≥2.
8. Those taking glucocorticoids.
9. Known hypersensitivity to anthracyclines, cyclophosphamide, taxanes, trastuzumab or pertuzumab.
10. Refuse contraception during treatment and within 8 weeks after completion of treatment for women of childbearing age.
11. Pregnant and lactating women.
12. After joining the test, a pregnancy test (+) before using the drug.
13. There are mental illness, cognitive impairment, unable to understand the test plan and side effects, unable to complete the test plan and follow-up workers (systematic evaluation is required before the trial is enrolled).
14. No personal freedom and independent civil capacity.
15. The investigator determined that the patient could not obtain long-term follow-up data (due to unavailability or serious concomitant diseases).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer patients
Enrollment: 159 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
The accuracy of carbon nanoparticle labelled lymph nodes in predicting axillary lymph nodes | 1-3 day before NST, the suspected lymph nodes will be injected carbon nanoparticle. During operation, carbon nanoparticle labelled lymph nodes will be identified and sent for examination.
  Before NST, one of the clinically assesed positive lymph nodes will be subjected to ultrasound-guided CNB or FNA, and a locating clip will be placed, meanwhile, a small amount of carbon nanoparticles suspension injection will be injected into or around the cortex of the locating lymph node and other clinically assessed positive lymph nodes. During operation, carbon nanoparticle labelled lymph nodes will be identified and sent for examination. Then calculate the accuracy of carbon nanoparticle labelled lymph nodes in predicting axillary lymph nodes for postoperative pathology.

SECONDARY OUTCOMES:
The consistency between the pre-operative FNA of clip labeled lymph nodes and post-operative pathology. | 1-3 day before NST, one of the cN+ nodes will be placed a locating clip. 1-3 days before surgery, the clip labeled node will be punctured again. During operation, the clip labeled node will be identified and sent for examination.
  Before NST, one of the clinically assesed positive lymph nodes will be subjected to ultrasound-guided CNB or FNA, and a locating clip will be placed. Before surgery, the clip labeled node will be punctured (FNA) again. During operation, the clip labeled node will be identified and sent for pathological examination. And then calculate the identification rate of labeled lymph nodes and the consistency between the pre-operative FNA of clip labeled lymph nodes and post-operative pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Zha, Doctor, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No